CLINICAL TRIAL: NCT02522949
Title: Evaluation of ColdZyme® Mouth Spray on Prevention and Alleviation of Induced Rhinovirus Upper Respiratory Tract Infection in Healthy Volunteers. A Double-blind, Randomized, Placebo-controlled Study
Brief Title: Evaluation of ColdZyme® Mouth Spray on Prevention and Alleviation of Rhinovirus Induced Common Cold
Acronym: COLDPREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymatica AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENZY-001
Record Dates: First submitted 2015-07-01; First posted 2015-08-13 (Estimated); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ColdZyme (Active Comparator): ColdZyme® mouth spray. Treatment (6 doses per day) will be applied for 11 days from the day of inoculation.
  Interventions: Device: ColdZyme® mouth spray
- Placebo (Placebo Comparator): Sugar based mouth spray manufactured to mimic ColdZyme® mouth spray. Treatment (6 doses per day) will be applied for 11 days from the day of inoculation.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: ColdZyme® mouth spray
  Arms: ColdZyme
Device: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the performance of ColdZyme® mouth spray on prevention and alleviation of induced rhinovirus upper respiratory tract infection in healthy volunteers. Half of participants will receive ColdZyme® mouth spray while the other half will receive placebo.

DETAILED DESCRIPTION:
Common colds can be caused by a number of viruses, e.g. rhinoviruses, coronaviruses, influenza viruses and others. The majority of colds are however caused by rhinovirus infection, which is responsible for up to 80% of all common colds. This study evaluates the effect of creating a physical barrier on the pharyngeal mucosal membrane to prevent or reduce virus cell entry during common cold infection to reduce total virus load and common cold symptoms in vivo in relation to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between 18-65 years. The investigator judges the definition of healthy by detailed medical history and physical examination.
2. Females of childbearing potential: should use reliable method of birth control. Reliable methods are hormonal contraceptives (combination pills, injections or implants), intrauterine device, condom or declared absence of sexual contact. Post-menopausal woman is defined as absence of menstrual discharge for at least two years.
3. Signed informed consent form prior to any study-related procedures.
4. Willingness and ability to complete the study.
5. Perceived to have had at least one cold per year.

Exclusion Criteria:

1. Smoker, during the last 12 months.
2. Any cold symptom within the last month such as sore throat, sneezing, rhinorrhoea, malaise, nasal obstruction or cough.
3. Presence of serum neutralising antibodies against human rhinovirus16 at screening.
4. Active allergic rhinitis, asthma or chronic obstructive pulmonary disease in last year.
5. Positive for fur allergy (if subject is likely to come in contact with the specific pet) and/or dust-mite allergy in skin prick test at screening.
6. Nasal disease, e.g. nasal polyposis, significant septal deviation, chronic rhinosinusitis, etc.
7. Females: Pregnant, breast-feeding or intentions to become pregnant during the study.
8. Active autoimmune disease in last year.
9. Evidence or history of drug or alcohol abuse.
10. Use of any prescribed or non-prescribed medication (except for contraceptives, paracetamol and ibuprofen) within 2 weeks prior to the first administration of investigational product until the end of study.
11. Use of any over the counter cold prophylaxis products such as C-vitamins, zinc or Echinacea within 1 month prior to the first administration of investigational product until the end of study.
12. Participation in other clinical study within 60 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Ahlström Emanuelsson, MD, Principal Investigator — Otorhinolaryngology, Skåne University Hospital, Lund.

REFERENCES:
- See also: Published article: A Randomized, Double-Blind, Placebo-Controlled Pilot Clinical Study on ColdZyme® Mouth Spray against Rhinovirus-Induced Common Cold — https://www.scirp.org/journal/paperinformation.aspx?paperid=79633

RESULTS

PARTICIPANT FLOW:
Groups:
- ColdZyme: ColdZyme® mouth spray. Treatment (6 doses per day) will be applied for 11 days from the day of inoculation.
  ColdZyme® mouth spray
- Placebo: Sugar based mouth spray manufactured to mimic ColdZyme® mouth spray. Treatment (6 doses per day) will be applied for 11 days from the day of inoculation.
  Placebo
Period: Overall Study
Arm/Group | ColdZyme | Placebo
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ColdZyme | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (5.7) | 23.3 (3.3) | 23.7 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  Sweden | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Viral Load in the URT
Description: Reduction in viral load in the URT(Upper Respiratory Tract), after challenge with rhinovirus, in relation to placebo
Time Frame: 7 days
Measure: Least Squares Mean (Standard Error); unit: log 10 copies/mL
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 23 | 23
log 10 copies/mL
  Oropharyngeal | 3.6 (0.6) | 3.3 (0.6)
  Nasal | 4.9 (0.6) | 4.1 (0.6)
Statistical Analysis 1: Comparison: ColdZyme vs Placebo; Oropharyngeal; Test type: Superiority; p = 0.7146, ANCOVA
Statistical Analysis 2: Comparison: ColdZyme vs Placebo; Nasal; Test type: Superiority; p = 0.3543, ANCOVA

2. Secondary Outcome: Prevention of Symptomatic URTI (Upper Respiratory Tract Infection)
Description: Reduction of number of days having a total symptom severity score of 6 or higher using a 5-graded Jackson scale, in relation to placebo.
  Will be assessed by the severity of cold symptoms quantified by the modified method of Jackson at peak day (day with highest score). A subject is considered to be a success if the total symptom score is below 6. Otherwise will the subject be classified as a failure to prevent symptomatic URTI.
Time Frame: 11 days
Measure: Count of Participants; unit: Participants
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  No (Success if total symptom score is below 6 on peak day) | 21 | 16
  Yes (Success if total symptom score is below 6 on peak day) | 2 | 7

3. Secondary Outcome: Prevention of Asymptomatic URTI
Description: Asymptomatic URTI will be assessed by quantification of viral load at peak day (day with highest viral load measured by oropharyngeal swab).
  Will be assessed by quantification of viral load at peak day (day with highest viral load). A subject is considered to be a success if the viral load is not different from the base-line value (from day 0). Otherwise will the subject be classified as a failure to prevent asymptomatic URTI.
Time Frame: 11 days
Measure: Count of Participants; unit: Participants
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 23 | 23
Participants
  No | 18 | 15
  Yes (success if viral load in oropharyngeal swab is 0 in peak day | 5 | 8

4. Secondary Outcome: Fewer Days With Symptomatic URTI
Description: The number of days with cold is defined as the sum of all days with a total score of ≥ 6 according to the modified method of Jackson.
Time Frame: 11 days
Measure: Median (Standard Deviation); unit: Days with symptomatic cold
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 23 | 23
Days with symptomatic cold | 2.0 (2.3) | 3.0 (3.1)

5. Secondary Outcome: Fewer Days With Asymptomatic URTI
Description: The number of days with asymptomatic URTI is defined as the sum of all days with a viral load significantly different from the baseline.
Time Frame: 11 days
Measure: Mean (Standard Deviation); unit: Days with asymptomatic cold
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 23 | 23
Days with asymptomatic cold | 1.0 (1.1) | 1.4 (1.0)

6. Secondary Outcome: Lower Level of Proinflammatory Proteins
Description: Nasal samples will be analysed for the quantity of IL-6 (Interleukin 6), IL-8 and IFNα (Interferon alpha).
Time Frame: 11 days
Measure: Mean (Standard Deviation); unit: pg*day/mL
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 23 | 23
pg*day/mL
  IL-6 | 273.93 (641.76) | 254.45 (494.69)
  IL-8 | 1863.36 (1597.92) | 2057.59 (1792.90)
  IFNα | 101.24 (66.65) | 101.15 (73.54)

7. Secondary Outcome: Lower Daily Total Symptom Score
Description: Jackson score was used and the *mean* sum of the score is reported. Jackson score is based on the sum of 5 severity points in the following scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 =very severe), where 0 is minimum and 4 is maximum score, for eight cold symptoms: sneezing, nasal obstruction, nasal discharge, sore throat, cough, headache, chilliness, and malaise.
Time Frame: Day 0-10
Measure: Least Squares Mean (Standard Error); unit: score on a 5 graded scale (0-4)
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 23 | 23
score on a 5 graded scale (0-4)
  Day 0 | 0.9 (0.3) | 0.2 (0.3)
  Day 1 | 1.5 (0.5) | 1.4 (0.5)
  Day 2 | 4.0 (0.8) | 4.3 (0.8)
  Day 3 | 4.6 (0.8) | 5.4 (0.8)
  Day 4 | 5.3 (0.8) | 5.5 (0.8)
  Day 5 | 4.3 (0.8) | 4.5 (0.8)
  Day 6 | 3.7 (0.7) | 3.7 (0.7)
  Day 7 | 3.3 (0.8) | 3.9 (0.8)
  Day 8 | 3.2 (0.9) | 3.3 (0.9)
  Day 9 | 3.0 (0.9) | 2.9 (0.9)
  Day 10 | 2.6 (0.9) | 3.1 (0.9)

8. Secondary Outcome: Lower Daily Score of Individual Symptoms
Description: Mean (average) value of the participants' score per symptom on day 10 is reported, i.e. per symptom, the total sum of participants self-reported Jackson score from 0 to 4, divided with number of participants on day 10.
  The Jackson scale for eight cold symptoms is used in the rating, using the following scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 =very severe , where 0 is no symptom and 4 is maximum symptoms (worsed), for eight cold symptoms: sneezing, nasal obstruction, nasal discharge, sore throat, cough, headache, chilliness, and malaise.
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 23 | 23
score on a scale
  Sneezing Day 10 | 0.22 (0.52) | 0.17 (0.65)
  Rhinorrhea Day 10 | 0.52 (0.85) | 0.57 (0.73)
  Nasal obstruction Day 10 | 0.39 (0.72) | 0.52 (0.85)
  Sore/scratchy throat Day 10 | 0.26 (0.62) | 0.30 (0.70)
  Cough Day 10 | 0.26 (0.69) | 0.65 (1.15)
  Headache Day 10 | 0.22 (0.67) | 0.13 (0.46)
  Malaise Day 10 | 0.48 (0.85) | 0.43 (0.73)
  Hoarseness Day 10 | 0.26 (0.54) | 0.30 (0.63)
  Chilliness Day 10 | 0.0 (0.0) | 0.4 (0.21)

9. Post Hoc Outcome: Area Under the Curve (AUC) for Day 3-10 in the Oropharyngeal Samples of Viral Load
Time Frame: Day 3, 4, 5, 7, 10
Population: Subjects with no viral load during the study excluded
Measure: Mean (Standard Deviation); unit: copies*day/mL
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 19 | 16
copies*day/mL | 6.6 (7.41) | 11.30 (6.17)
Statistical Analysis 1: Comparison: ColdZyme vs Placebo; Test type: Other; p = 0.0232, Exact Wilcoxon rank sum test

10. Post Hoc Outcome: Number of Days With Asymptomatic Cold (Oropharyngeal Sample)
Time Frame: 11 days
Population: Subjects with no viral load during the study excluded
Measure: Median (Standard Deviation); unit: Days with asymptomatic cold
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 19 | 16
Days with asymptomatic cold | 1.0 (1.0) | 2.0 (1.0)

11. Post Hoc Outcome: Number of Days With Asymptomatic Cold (Nasal Sample)
Time Frame: 11 days
Population: Subjects with no viral load during the study excluded
Measure: Mean (Standard Deviation); unit: Days with asymptomatic cold
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 19 | 16
Days with asymptomatic cold | 3.0 (1.5) | 4.0 (1.5)

12. Post Hoc Outcome: Number of Days With Symptomatic Cold
Time Frame: 11 days
Population: Subjects with no symptomatic cold during the study excluded
Measure: Median (Standard Deviation); unit: Days with symptomatic cold
Arm/Group | ColdZyme | Placebo
Number analyzed (Participants) | 21 | 16
Days with symptomatic cold | 3.0 (2.1) | 6.5 (2.7)

ADVERSE EVENTS:
Arm/Group | ColdZyme | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 3/23 | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ColdZyme (N=23) | Placebo (N=23)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (3)
Enlarged uvula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the small sample size and the low infection rate of 76% and the power calculation being based on an estimated infection rate of >85%, exploratory analyses of subjects who experienced an infection (subjects with a value of viral load above 0 in pharyngeal or nasal sample any time during the study period) were performed. Peak viral load turned out to be an unreliable parameter with sometimes two peaks for the same subject. Thus, viral load as AUC was analyzed in the post hoc analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No